CLINICAL TRIAL: NCT05097482
Title: Triceps Surae Muscle Characteristics in Hemiparetic Stroke Survivors: Clinical Implications From Ultrasonographic Evaluation
Brief Title: Triceps Surae Ultrasonographic Characteristics in Hemiparetic Stroke Survivors
Acronym: TriUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alessio Baricich (Other)
Responsible Party: Sponsor-Investigator, Alessio Baricich, Professor in Physical and Rehabilitation Medicine, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Organization: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Other Study IDs: TriUS
Record Dates: First submitted 2021-08-31; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Spastic Foot; Stroke
Keywords: post-stroke spasticity; muscle; ultrasound
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate, in hemiparetic patients, changes in muscle ultrasound structure about the focal treatment of spasticity with botulinum toxin type A. For this purpose, the analysis of the mean echo intensity will be carried out on ultrasound acquisitions, identifying the possible correlations between the muscle echogenicity, the variations in the pennation angle, and the length of the fascicles.

For image processing operations, ImageJ software was applied.

ELIGIBILITY:
Inclusion Criteria:

* unilateral ischaemic or haemorrhagic stroke (documented with clinical examination and neuroradiological findings)
* presence of spasticity at lower limb muscles, at least grade 1+ in the modified Ashworth Scale 3.
* age ≥ 18 years

Exclusion Criteria:

* inability to walk before stroke
* presence of severe cognitive impairment
* presence of other musculoskeletal, neurological or cardiopulmonary impairment which can interfere with clinical findings
* presence of skin lesions that can contraindicate BoNT-A treatment
* previous surgical myotendinous elongation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects already treated for focal post-stroke spasticity in our Unit
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-12-13 (Estimated); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
muscle structure variations | single measure through study completion (1 year)
  The primary outcome consists in detecting muscle structure variations during the procedure.
  This measure will be related to the time frame between the first inoculation and the moment of image acquisition, and to the number of therapeutic cycles performed. The aim is to determine the potential correlation between BoNT-A injection and muscle structure evolution.
  The time point of assessment is not pre-defined but the time since stroke onset and, if applicable, from the first BoNT-A injection will be recorded.
  Each participant will be assessed once during the overall duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore della Carità University Hospital, Novara, Italy